CLINICAL TRIAL: NCT02707874
Title: Comparing the Delivery of Local Anesthetic by Programmed Intermittent Bolus Versus Continuous Infusion Through a Popliteal Sciatic Nerve Catheter for Analgesia Following Major Ankle Surgery
Brief Title: PIB Versus CI Through a Popliteal Sciatic Nerve Catheter for Analgesia Following Major Ankle Surgery
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REB#13-6466
Record Dates: First submitted 2015-11-20; First posted 2016-03-14 (Estimated); Last update posted 2016-10-31 (Estimated); Status verified 2016-10

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative | interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- CI 0.2% ropivacaine (Active Comparator): Patients in Group Continuous Infusion (CI) will receive continuous infusion of 0.2% ropivacaine at 5 mL/hour; total 4-hourly consumption = 20 mL = 40 mg ropivacaine.
  • All patients will be able to self-administer PCA boluses of 5 mL of ropivacaine 0.2% at intervals of 30 minutes as required.
  2) Oral patient controlled analgesia (PCA) using oxycodone or hydromorphone. Patients under 70 years of age will receive either 10 mg of oxycodone or 2 mg of hydromorphone 2 hourly as needed, and patients 70 years of age or older will receive 5 mg of oxycodone or 1 mg of hydromorphone 2 hourly as needed.
  3) Oral acetaminophen 1,000 mg 6 hourly.
  Interventions: Drug: CI 0.2% ropivacaine
- PIB 0.2% ropivacaine (Active Comparator): Patients in Group programmed intermittent boluses (PIB) will receive automated programmed intermittent boluses of 10 mL of ropivacaine 0.2% every 2 hours; total 4-hourly consumption = 20 mL = 40 mg ropivacaine.
  • All patients will be able to self-administer PCA boluses of 5 mL of ropivacaine 0.2% at intervals of 30 minutes as required.
  2) Oral patient controlled analgesia (PCA) using oxycodone or hydromorphone. Patients under 70 years of age will receive either 10 mg of oxycodone or 2 mg of hydromorphone 2 hourly as needed, and patients 70 years of age or older will receive 5 mg of oxycodone or 1 mg of hydromorphone 2 hourly as needed.
  3) Oral acetaminophen 1,000 mg 6 hourly.
  Interventions: Drug: PIB 0.2% ropivacaine

INTERVENTIONS:
Drug: CI 0.2% ropivacaine — Patients in Group CI will receive continuous infusion of 0.2% ropivacaine at 5 mL/hour; total 4-hourly consumption = 20 mL = 40 mg ropivacaine. All patients will be able to self-administer PCA boluses of 5 mL of ropivacaine 0.2% at intervals of 30 minutes as required
  Other Names: ropivacaine 0.2% Continuous infusion
  Arms: CI 0.2% ropivacaine
Drug: PIB 0.2% ropivacaine — Patients in Group Programmed intermittent bolus (PIB) will receive automated programmed intermittent boluses of 10 mL of ropivacaine 0.2% every 2 hours; total 4-hourly consumption = 20 mL = 40 mg ropivacaine. All patients will be able to self-administer PCA boluses of 5 mL of ropivacaine 0.2% at intervals of 30 minutes as required
  Other Names: ropivacaine 0.2% Programmed intermittent bolus
  Arms: PIB 0.2% ropivacaine

SUMMARY:
This is a clinical study to investigate and compare a new programmed intermittent bolus (PIB) delivery method for continuous popliteal sciatic nerve block for pain relief in patients undergoing major ankle surgery compared with the current practice of continuous local anesthetic infusion (CI).

DETAILED DESCRIPTION:
Peripheral nerve blocks are commonly used for upper and lower limb surgery. Continuous popliteal sciatic nerve block achieved by delivery of local anesthetic through a perineural catheter plays an important role in post-operative pain control after major orthopedic surgeries of the ankle and foot. Factors affecting the success and clinical outcome of continuous sciatic nerve blocks include the accuracy of catheter placement, the local anesthetic dose (volume and concentration), and the infusion method.

Methods of local anesthetic infusion commonly used for peripheral nerve blockade include continuous infusion (CI) and CI combined with patient-controlled analgesic (PCA) boluses. A third option, regular intermittent boluses of local anesthetic, is not commonly used as it usually requires manual administration by a healthcare provider and is thus time and labor-intensive. Recently, however, infusion pumps capable of providing automated programmed intermittent bolus (PIB) dosing have become available.

The premise of PIB dosing is that it results in more extensive spread of local anesthetic around nerves, and thus more effective sensory block and analgesia. PIB dosing regimens have been extensively studied in labor epidural analgesia, where they have been shown to decrease local anesthetic consumption and improve maternal satisfaction when compared with continuous infusion regimens.

In contrast, there has been little investigation into PIB dosing regimens in the context of continuous peripheral nerve blockade. In 2005, Taboada et al 2 published a study that compared automated PIB dosing with CI dosing of local anesthetic for continuous popliteal sciatic nerve blockade. In both regimens, patients were also allowed to administer PCA boluses of local anesthetic as needed to improve the quality of the nerve block. The authors found that the automated PIB dosing regimen resulted in patients using less local anesthetic and fewer PCA boluses, while providing equivalent analgesia. There was a non-significant trend to lower pain scores in the PIB group of patients. These effects are attributed to better perineural spread of local anesthetic with the PIB regimen. No other studies have been conducted to confirm these benefits.

The reduced local anesthetic requirement is of particular advantage in patients who are discharged home with a nerve block catheter in situ as the supplied reservoir of local anesthetic will last longer. Ambulatory infusion pumps with both PIB and PCA features are now commercially available. The investigators hypothesize that a PIB+PCA dosing regimen using one of these new ambulatory infusion pumps will provide more effective postoperative analgesia with less local anesthetic consumption than the CI+PCA dosing regimen.

ELIGIBILITY:
Inclusion Criteria:

* Inpatients having major foot and ankle surgery that will benefit from continuous popliteal sciatic nerve block with an indwelling catheter
* American Society Anesthesiologists (ASA) physical status I-III
* 18-85 years of age, inclusive
* 40-120 kg, inclusive
* 150 cm of height or greater

Exclusion Criteria:

* Patients who undergo iliac crest bone graft harvesting as part of their surgery
* Preexisting neurological deficits or peripheral neuropathy in the distribution of the sciatic nerve
* Local infection
* Contraindication to regional anesthesia e.g. bleeding diathesis, coagulopathy
* Chronic pain disorders
* History of use of over 30mg oxycodone or equivalent per day
* Allergy to local anesthetics
* History of significant psychiatric conditions that may affect patient assessment
* Pregnancy
* Inability to provide informed consent

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2014-10; Primary Completion 2017-12 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Average numerical rating score (NRS) for pain | post-operative 48 hours

SECONDARY OUTCOMES:
NRS for pain at rest and with movement at specified time points | post-operative 48 hours
Number of local anesthetic PCA boluses administered | post-operative 48 hours
Total dose of local anesthetic | post-operative 48 hours
Patient satisfaction, on a 0-10 NRS | post-operative 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Ki Jinn Chin, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- Toronto Western Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
by publication

REFERENCES:
- [Background] George RB, Allen TK, Habib AS. Intermittent epidural bolus compared with continuous epidural infusions for labor analgesia: a systematic review and meta-analysis. Anesth Analg. 2013 Jan;116(1):133-44. doi: 10.1213/ANE.0b013e3182713b26. Epub 2012 Dec 7. PMID 23223119
- [Background] Taboada M, Rodriguez J, Bermudez M, Amor M, Ulloa B, Aneiros F, Sebate S, Cortes J, Alvarez J, Atanassoff PG. Comparison of continuous infusion versus automated bolus for postoperative patient-controlled analgesia with popliteal sciatic nerve catheters. Anesthesiology. 2009 Jan;110(1):150-4. doi: 10.1097/ALN.0b013e318191693a. PMID 19104182
- [Background] Chludzinski A, Irani C, Mascha EJ, Kurz A, Devereaux PJ, Sessler DI. Protocol understanding and anxiety in perioperative clinical trial patients approached for consent on the day of surgery. Mayo Clin Proc. 2013 May;88(5):446-54. doi: 10.1016/j.mayocp.2012.12.014. PMID 23639498
- [Derived] Short AJ, Ghosh M, Jin R, Chan VWS, Chin KJ. Intermittent bolus versus continuous infusion popliteal sciatic nerve block following major foot and ankle surgery: a prospective randomized comparison. Reg Anesth Pain Med. 2019 Sep 29:rapm-2018-100301. doi: 10.1136/rapm-2018-100301. Online ahead of print. PMID 31570495